CLINICAL TRIAL: NCT04306055
Title: Blood Donor Recruitment During Epidemic of COVID-19 in Guangzhou, China
Brief Title: Blood Donor Recruitment During Epidemic of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Principal Investigator, OUYANG Jian, Investigator, Guangzhou Blood Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Blood donor recruitment
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Blood Donation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Questionnaire with precaution information (Experimental): Questionnaire in this group includes information about precaution of blood donation during epidemic of COVID-19.
  Interventions: Other: Questionnaire with precaution information
- Questionnaire without precaution information (Experimental): Questionnaire in this group dose not include information about precaution of blood donation during epidemic of COVID-19.
  Interventions: Other: Experimental: Questionnaire without precaution information
- No questionnaire group (No Intervention): Ever donors in this group would not receive the questionnaire.

INTERVENTIONS:
Other: Questionnaire with precaution information — Ever blood donors in this group would receive a questionnaire which includes some information about how donors can donate safely and how blood center will protect the blood donors during the epidemic of COVID-19.
  Arms: Questionnaire with precaution information
Other: Experimental: Questionnaire without precaution information — Ever blood donors in this group would receive a questionnaire which dose not include the information above.
  Arms: Questionnaire without precaution information

SUMMARY:
In December 2019, an unknown pneumonia rapidly spread in Wuhan, China, a new coronavirus, 2019 novel coronavirus (2019-nCoV), aroused the attention of the entire world. On January 31, 2020, World Health Organization (WHO) announced the outbreak of Coronavirus Disease 2019 (COVID-19) in China as a Public Health Emergency of International Concern. The number of volunteer non-remunerated blood donors decreased because of quarantine, caring for relatives, and fear of exposure to COVID-19. Due to the blood shortage, patient blood management and cessation of elective surgery are contributing to decreased demand, but sepsis may increase requirements and significant reductions will not be possible in areas such as trauma, cancer patients, hereditary haemolytic anaemias and childbirth. Therefore, recruiting enough blood donors during the epidemic is vital for public health in China, and also worldwide. In order to assess the effects of a questionnaire on blood donor recruitment, the investigators designed two kinds of self-administered, standardized and structured questionnaires. In addition of the basic socio-demographic characteristics, one questionnaire includes the information of precautions of blood donation during epidemic, and the other dose not. The questionnaires were randomly sent to ever blood donors, and the same number of ever blood donors are coded as control.

DETAILED DESCRIPTION:
In order to assess the effects of a questionnaire on blood donor recruitment, the investigators designed two kinds of self-administered, standardized and structured questionnaires. In addition of the basic socio-demographic characteristics, one questionnaire includes the information of precautions of blood donation during epidemic, and the other dose not.

Information of precautions of blood donation during epidemic included taking donor's temperature and enhancing hand disinfection before donation etc.

The questionnaires were randomly sent to ever blood donors, and at the same day, equal number of ever blood donors as the ones who filled the questionnaire are coded as control.

ELIGIBILITY:
Inclusion Criteria:

* Blood donors whose last donation were between 1 Feb to 31 March, 2019.

Exclusion Criteria:

* Blood donors whose blood test results were positive. Blood donors who were aged above 60. Blood donors whose cell phone number was obviously invalid.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19491 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Differences of attitude about blood donation towards different questionnaires | 1 day
  Compare participants' intention of blood donation after they read different information in the questionnaire.

SECONDARY OUTCOMES:
Rates of blood donation during 3 weeks | 3 weeks
  Blood donation rate of 3 groups will be followed

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No